CLINICAL TRIAL: NCT05869318
Title: RESEC: Respiratory Effects of E-Cigarettes in Obese Youth
Brief Title: Respiratory Effects of E-Cigarettes in Obese Youth
Acronym: RESEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Dharini Bhammar, Assistant Professor, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-22219; NCI-2023-04458 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: E-Cig Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaping (Experimental): All participants will undergo two vaping sessions: one using their own device and one using the study device
  Interventions: Other: ECIG own; Other: ECIG Vuse

INTERVENTIONS:
Other: ECIG own — Participants will vape using their own ecig device
Other: ECIG Vuse — Participants will vape a VUSE e-cigarette (GOLD 5%)

SUMMARY:
To determine vaping behaviors and respiratory function in obese and nonobese youth e-cigarette users.

DETAILED DESCRIPTION:
The investigators hypothesize that obese youth e-cigarette users will have increased e-cigarette use that will worsen respiratory function. The approach will involve a clinical trial where vaping behaviors (using puff topography) and respiratory function (spirometry, plethysmography, and diffusion capacity) will be assessed while participants vape with their own e-cigarette and, on a separate visit, with the VUSE e-cigarette.

ELIGIBILITY:
Inclusion Criteria:

* a current e-cigarette user (≥1 vaping bout daily) for at least the past 3 months,
* 21-25 years old,
* willing to abstain from all tobacco and nicotine for at least 12 hours prior to lab sessions,
* willing to complete five lab visits lasting up to 4 hours each,
* able to read and speak English,
* willing to provide informed consent.

Exclusion Criteria:

* self-reported diagnosis of lung disease including asthma or cystic fibrosis
* history of cardiac event or distress within the past 3 months
* history of metabolic disease including thyroid disease or diabetes
* history of orthopedic or neuromuscular problems that preclude exercise
* currently pregnant (determined using urine pregnancy test), planning to become pregnant, delivered a child in the past 6 weeks even if not breastfeeding, or currently breastfeeding
* use of other tobacco products >10 days in the past month
* current marijuana use >10 times per month
* currently engaging in a vaping cessation attempt
* ) competitive athlete or individual currently engaged in an exercise training program involving 420min or more (moderate intensity aerobic activity) or 210 min or more (vigorous intensity aerobic activity) per week with the goal of participating in a competitive event or marathon, triathlon, etc. Participants who are engaged in usual physical activity (e.g., walking dog, biking to work, etc.) but not engaged in a "structured exercise training program" will not be excluded.
* plans to leave the Columbus or central Ohio region within the next year.

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second | Change from 0 to 35 minutes
  Spirometry will be completed before and after a 35 min vaping session
Functional residual capacity | Change from 0 to 35 minutes
  Plethymosgraphy will be completed before and after a 35 min vaping session
Diffusion capacity | Change from 0 to 35 minutes
  DLCO will be completed before and after a 35 min vaping session
Airway resistance | Change from 0 to 35 minutes
  Plethymosgraphy to measure airway resistance (Raw) will be completed before and after a 35 min vaping session
Puff count | 35 minutes
  E-cig puff topography data collection for abuse liability
Average Puff duration | 35 minutes
  E-cig puff topography data collection for abuse liability
Average Puff volume | 35 minutes
  E-cig puff topography data collection for abuse liability

SECONDARY OUTCOMES:
Tiffany-Drobes Questionnaire of Smoking Urges | Change from 0 to 35 minutes
  Assess E-cig craving/suppression of craving
Respiratory health questionnaire | Change from 0 to 35 minutes
  Assess respiratory symptoms
Exhaled carbon monoxide | Change from 0 to 35 minutes
  Assess carbon monoxide in exhaled air

CONTACTS AND LOCATIONS:
Overall Officials: Dharini M Bhammar, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT05869318/ICF_001.pdf